CLINICAL TRIAL: NCT06036797
Title: Efficacy and Safety of Hydromorphone-ropivacaine Versus Sufentanil-ropivacaine for Epidural Labor Analgesia: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Hydromorphone-ropivacaine Versus Sufentanil-ropivacaine for Epidural Labor Analgesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCHH_003
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Analgesia; Labor Pain
MeSH Terms: conditions — Agnosia; Labor Pain | interventions — Hydromorphone; Sufentanil; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Group 1 will be administered with 15 ug/ml hydromorphone and 0.08% ropivacaine
  Interventions: Drug: Hydromorphone; Drug: Ropivacaine
- Group 2 (Experimental): Group 2 will be administered with 17.5 ug/ml hydromorphone and 0.08% ropivacaine
  Interventions: Drug: Hydromorphone; Drug: Ropivacaine
- Group 3 (Experimental): Group 3 will be administered with 20 ug/ml hydromorphone and 0.08% ropivacaine
  Interventions: Drug: Hydromorphone; Drug: Ropivacaine
- Group 4 (Active Comparator): Group 4 will be administered with 0.4 ug/ml sufentanil and 0.08% ropivacaine
  Interventions: Drug: Sufentanil; Drug: Ropivacaine

INTERVENTIONS:
Drug: Hydromorphone — For those in Group 1 : they will be administered with 15 ug/ml hydromorphone, For those in Group 2 : they will be administered with 17.5 ug/ml hydromorphone, For those in Group 3 : they will be administered with 20 ug/ml hydromorphone
  Arms: Group 1; Group 2; Group 3
Drug: Sufentanil — For those in Group 4 : they will be administered with 0.4 ug/ml sufentanil
  Arms: Group 4
Drug: Ropivacaine — 0.08% ropivacaine will be co-administrated for epidural labor analgesia in four arms

SUMMARY:
The purpose of this study is to compare the effects of three different doses of hydromorphone combined with ropivacaine and sufentanil combined with ropivacaine in epidural labor analgesia through prospective clinical trials, so as to explore whether hydromorphone combined with ropivacaine has advantages in epidural labor analgesia, and find out the optimal dose of hydromorphone.

Participants will be randomly allocated to four groups : Group 1, Group 2, Group 3 and Group 4. For those in Group 1 : they will be administered with 15 ug/ml hydromorphone and 0.08% ropivacaine for epidural labor analgesia, For those in Group 2 : they will be administered with17.5 ug/ml hydromorphone and 0.08% ropivacaine for epidural labor analgesia, For those in Group 3 : they will be administered with 20 ug/ml hydromorphone and 0.08% ropivacaine for epidural labor analgesia, For those in Group 4 : they will be administered with 0.4 ug/ml sufentanil and 0.08% ropivacaine for epidural labor analgesia.

The goal of this clinical trial is to provide a new treatment option for pregnant women in epidural labor analgesia, and to provide a basis for hydromorphone combined with ropivacaine in epidural labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II
* a single fetus
* competent to provide informed consent

Exclusion Criteria:

* severe respiratory diseases including hypoxemia, respiratory failure and severe pneumonia
* severe circulatory diseases including acute decompensated heart failure and peripartum cardiomyopathy
* placenta previa

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-09-17 (Actual); Primary Completion 2023-10-17 (Estimated); Study Completion 2023-10-17 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | 30 minutes-1 hour
  VAS will be monitored and recorded at 6 time points, including the time of entering the operating room(Time 0), when the first dose is given for 5 minutes(Time 1), when the first dose is given for 15 minutes(Time 2), when the first dose is given for 30 minutes(Time 3), 30 minutes after delivery (Time 4), and 60 minutes after delivery (Time 5). The VAS consists of a 10 cm line, with two end points representing 0 (no pain) and 10 (pain as bad as it could possibly be).

SECONDARY OUTCOMES:
Heart rate(HR) | 30 minutes-1.5 hours
  HR will be monitored and recorded at 5 time points, including the time of entering the operating room(Time 0),when the first dose is given for 5 minutes(Time 1), when the first dose is given for 15 minutes(Time 2), 30 minutes after delivery (Time 3), and 60 minutes after delivery (Time 4).
Mean arterial pressure(MAP) | 30 minutes-1.5 hours
  MAP will be monitored and recorded at 5 time points, including the time of entering the operating room(Time 0),when the first dose is given for 5 minutes(Time 1), when the first dose is given for 15 minutes(Time 2), 30 minutes after delivery (Time 3), and 60 minutes after delivery (Time 4).
Pulse oxygen saturation | 30 minutes-1.5 hours
  Pulse oxygen saturation will be monitored and recorded at 5 time points, including the time of entering the operating room(Time 0),when the first dose is given for 5 minutes(Time 1), when the first dose is given for 15 minutes(Time 2), 30 minutes after delivery (Time 3), and 60 minutes after delivery (Time 4).
Duration of analgesia | 30 minutes-1.5 hours
  Defined as the time from labor analgesia to delivery of the fetus.
The number of compressions | 30 minutes-1.5 hours
  The number of compressions by electronic analgesia pump from labor analgesia to delivery of the fetus.
Adverse reactions | 30 minutes-1.5 hours
  The occurrence of adverse reactions(nausea, vomiting, skin itching and other adverse reactions).
The Apgar scores | 1 minute and 5 minutes after birth
  The Apgar scores of 1 minute and 5 minutes after birth will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China